CLINICAL TRIAL: NCT05015244
Title: Impact of Von Willebrand Factor-platelet Aggregates in Patients With Type 2B Disease
Acronym: Von2B
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2018-A03005-50
Record Dates: First submitted 2021-07-20; First posted 2021-08-20 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2021-08

CONDITIONS: Von Willebrand Disease, Type 2B
Keywords: VWF; Type 2B von willebrand disease
MeSH Terms: conditions — von Willebrand Disease, Type 2 | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Von Willebrand Disease Type 2B patient with neurological symptoms (Experimental): evaluation of patients using 3T (Tesla) Magnetic Resonance Imaging (MRI) and series of neuropsychological tests that cover virtually all cognitive domains.
  Interventions: Procedure: 3T (Tesla) Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Procedure: 3T (Tesla) Magnetic Resonance Imaging (MRI) — Neurological evaluation using MRI and neuropsychological tests
  Other Names: Series of neuropsychological tests that cover virtually all cognitive domains

SUMMARY:
The working hypothesis is that patients with Von Willebrand Disease-type 2B may have neurological symptoms due to the chronic formation of platelets/Von Willebrand Factor aggregates. Interestingly, several patients present nonspecific neurological symptoms (nystagmus, headaches, memory disorder, …) which may be associated with cerebral microangiopathy and chronic microvessel inflammation secondary to Von Willebrand Disease-type 2B due to chronic exposure to Von Willebrand Factor-platelets complexes.

DETAILED DESCRIPTION:
Investigator will use an extensive series of neuropsychological tests that cover virtually all cognitive domains. A measurement of global cognitive function will be assessed by the Mini Mental State Examination (MMSE). The verbal memory function will be assessed by the Rey Auditory Verbal Learning Test (RAVLT). Visuospatial memory will be administered by the Rey's Complex Figure Test (RCFT). To evaluate speed of mental processes, Stroop test (three subtasks), the Paper and Pencil Memory Scanning Task (four subtasks), the Symbol-Digit Substitution Task will be used. To evaluate attention, the verbal series attention test (VSAT) will be used. To register subjective cognitive failures investigator will administer the Cognitive failures questionnaire (CFQ). The neurological evaluation will be completed with 3T (Tesla) Magnetic Resonance Imaging (MRI) with different MRI sequences including T1 3D SPACE, FLAIR 3D , 3D SWI (Susceptibility weighted imaging) and 2D EPI (Echo Planar Imaging) to address the presence of cerebral small vessel disease. The presence of each of the four MRI markers for cerebral small vessel disease (white matter hyperintensities, lacunes, cerebral microbleeds and perivascular spaces will be addressed.

ELIGIBILITY:
Inclusion Criteria:

* patients with type 2B disease
* neurological signs
* signature of inform consent

Exclusion Criteria:

* contraindication for MRI
* Pregnant women
* other hemorrhagic disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Rate of cerebral lesions in patients with type 2B disease | at the inclusion
  Analysis of MRI sequences and % of patients with cerebral lesions

SECONDARY OUTCOMES:
Global cognitive function evaluation | at the inclusion
  Mini Mental State Examination (MMSE) will be used
Verbal memory function evaluation | at the inclusion
  Rey Auditory Verbal Learning Test (RAVLT) will be used
Visuospatial memory evaluation | at the inclusion
  Rey's Complex Figure Test (RCFT) will be used
Speed of mental processes evaluation | at the inclusion
  Stroop test will be used
Attention evaluation | at the inclusion
  Verbal series attention test (VSAT) will be used
Subjective cognitive failures evaluation | at the inclusion
  Cognitive failures questionnaire (CFQ) will be used

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Caen, Calvados, France

IPD SHARING:
Plan to Share IPD: Undecided